CLINICAL TRIAL: NCT00779740
Title: Clinical Equivalency Study of Two Formulations of Mometasone Furoate Nasal Spray
Brief Title: Equivalency Study of Two Formulations of Mometasone Furoate Nasal Spray (Study P04419)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04419; JPC-04-342-41
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Formulation Group (Experimental)
  Interventions: Drug: mometasone furoate
- Old Formulation Group (Active Comparator)
  Interventions: Drug: mometasone furoate

INTERVENTIONS:
Drug: mometasone furoate — The dose will be 50 mcg as MF in one spray (100 µL) per nostril two times a day (morning and night) for 2 weeks. The daily dose of MF will be 200 mcg.
  Other Names: Nasonex; SCH 32088
  Arms: New Formulation Group
Drug: mometasone furoate — The dose will be 50 mcg as MF in one spray (50 µL) per nostril two times a day (morning and night) for 2 weeks. The daily dose of MF will be 200 mcg.
  Other Names: Nasonex; SCH 32088
  Arms: Old Formulation Group

SUMMARY:
This is a multicenter, open-label, randomized, parallel group comparison study to verify the clinical equivalency of the old formulation (50 mcg as mometasone furoate [MF] in 50 μL of solution per spray) to the new formulation (50 mcg as MF in 100 μL of solution per spray) in patients with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of mongoloid race residing in Japan who satisfy all of the following criteria:

  * Patients having symptoms of perennial allergic rhinitis of moderate or severe degree, according to the classification of severity in the guidelines for the treatment of nasal allergy (partial revision) as well as a score of at least 4 in the score of 4 nasal symptoms, at the time of obtaining informed consent and during the pretreatment observation period.
  * Patients with a positive skin reaction test or specific IgE antibody quantitation, and with a positive cytological examination of nasal discharge (eosinophils) or nasal challenge test.
  * Outpatients who are at least 16 years of age at the time of informed consent obtained.
  * Male or female.
  * Patients who have the ability to give written informed consent (informed consent of the guardian must also be obtained for patients younger than 20 years).
  * Patients who can keep nasal allergy diary without fail.

Exclusion Criteria:

* Patients with coexisting tuberculous disease or lower respiratory tract infection, or patients who, at the time of registration, have acute upper respiratory tract infection, acute pharyngitis, acute amygdalitis etc.
* Patients with coexisting infections or systemic mycosis for which there are no effective antibiotics.
* Patients with unhealed nasal septum ulcers, nasal surgery scar, or nasal trauma.
* Patients with a history of hypersensitivity to steroids or mometasone furoate.
* Patients who are pregnant or nursing or who may be pregnant and patients or patients' partners who desire to become pregnant during the study period.
* Patients with severe hepatic, renal, cardiac, hematological disease, diabetes mellitus, hypertension or other serious coexisting diseases and whose general condition is poor.
* Patients also allergic to pollen and the pollen release season occurs during the study period.
* Patients with vasomotor rhinitis or eosinophilic rhinitis.
* Patients with a nasal condition which may interfere with efficacy evaluation of the investigational product.
* Patients who develop disease affecting nasal symptoms during the pretreatment observation period, i.e., during the 7 days before actual registration.
* Patients who are participating or have participated in a clinical trial of another investigational drug within 120 days (4 months) before the day of the informed consent for this study.
* Patients for whom the period of discontinuation of previous treatment effective for allergic rhinitis before the start of the investigational product administration is not sufficient or who cannot avoid its use.
* Patients receiving specific desensitization therapy or nonspecific modulation therapy or who had just discontinued such therapies within 90 days (3 months) before providing consent to this study (unless such therapies are ongoing as maintenance therapy and had been started 180 days [6 months] or more before consent to this study).
* Other patients judged inappropriate for study by the investigator or subinvestigator.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-02-01 (Actual); Primary Completion 2005-04-01 (Actual); Study Completion 2005-04-01 (Actual)

PRIMARY OUTCOMES:
Change in 4 nasal symptom score (sneezing attack, rhinorrhea, nasal congestion, and nasal itching) from baseline at Week 2. | After 2 weeks of treatment

SECONDARY OUTCOMES:
Change in each nasal symptom (sneezing attack, rhinorrhea, nasal congestion, and nasal itching). | After 2 weeks of treatment
Overall improvement | 2 weeks
Adverse events | From initial day of treatment until treatment is stopped.
Laboratory tests | At 7 or more days before treatment start, and after 2 weeks of treatment

REFERENCES:
- [Result] T. Ishikawa et. al; Practica otologica. Suppl.123 Page1-18 (2008.12) -Japanese language journal